CLINICAL TRIAL: NCT01033032
Title: Phase I/II Trial of Amrubicin as Second- or Third-Line Treatment for Patients With HER2-Negative Metastatic Breast Cancer
Brief Title: Trial of Amrubicin as Treatment for Patients With HER2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 161
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Amrubicin
MeSH Terms: conditions — Breast Neoplasms | interventions — amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amrubicin Phase I/II (Experimental): Systemic therapy with amrubicin
  Interventions: Drug: Amrubicin

INTERVENTIONS:
Drug: Amrubicin — Phase I: dose-escalating portion with the starting dose of amrubicin at 90mg/m^2 IV q21 days. Dose escalations are as follows:
  DL2 - 100mg/m^2; DL3 - 110mg/m^2; and DL4 - 120mg/m^2. All cycles are q21 days
  Phase II: Amrubicin will be administered at the maximum tolerated dose established in Phase I by IV every 21 days
  Other Names: Systemic therapy

SUMMARY:
Doxorubicin has been an integral part of the treatment of women with breast cancer for many years. Since amrubicin may have more activity than doxorubicin, as well as less cardiotoxicity, evaluation of amrubicin in the treatment of advanced breast cancer should be a priority. In this Phase II study, the investigators propose an evaluation of single-agent amrubicin as second- or third-line treatment for women with metastatic breast cancer.

DETAILED DESCRIPTION:
This will be a phase I/II study where phase I will evaluate the maximum tolerated dose of amrubicin, and phase II will assess the progression free survival of patients with HER2-negative metastatic breast cancer using the dose established in the phase I portion.

ELIGIBILITY:
Inclusion Criteria:

1. Females >=18 years of age.
2. Histologic diagnosis of HER2-negative breast cancer. HER-2 negativity must be confirmed by one of the following:

   * FISH-negative (FISH ratio <2.2), or
   * IHC 0-1+, or
   * IHC 2-3+ AND FISH-negative (FISH ratio <2.2)
3. Evidence of metastatic or locally advanced, inoperable breast cancer.
4. Minimum of 1 and maximum of 2 prior metastatic breast cancer chemotherapy regimens.
5. Patients with prior anthracycline therapy are eligible, provided their previous anthracycline was ≥6 months prior to study entry.
6. Measurable disease per RECIST criteria version 1.1
7. Left ventricular ejection fraction (LVEF) ³50% by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA).
8. Patients must have QTc interval of <=450 msec.
9. No intercurrent significant medical conditions or cardiac illness.
10. Patients must be >=3 weeks since last chemotherapy, and recovered from all acute toxicities, with the exception of alopecia.
11. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2.
12. Adequate organ function including the following:

    * ANC >=1500 cells/mL
    * Platelet count >=100,000 cells/mL
    * Hemoglobin >=9 g/dL
    * Total bilirubin <=1.5 x ULN; AST/ALT <=2.5 x ULN, (except if due to hepatic metastases, then <=5 x ULN)
    * Serum creatinine <1.5 x ULN
13. Women of childbearing potential must have a negative serum or urine pregnancy test performed <=7 days prior to start of treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
14. Patients must be accessible for treatment and follow-up.
15. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.
16. Patients who are on anticoagulation are acceptable if the therapeutic anticoagulation is stable. Additionally, the patient's INR must be adequate if the patient is receiving treatment with coumadin.
17. Prior hormonal therapy for metastatic breast cancer is permitted; however, the therapy must be discontinued prior to the patient's enrollment in this study.

Exclusion Criteria:

1. Any concurrent therapy with other investigational, chemotherapeutic, or hormonal therapy.
2. Prior treatment with >=3 regimens of cytotoxic therapy in the advanced disease setting. (Any number of previous hormonal therapies are acceptable, as long as the therapy is discontinued prior to the patient's enrollment into this study).
3. Major surgery or systemic therapy <=3 weeks of study treatment.
4. Prior high-dose chemotherapy requiring hematopoietic stem cell support.
5. Prior radiation therapy to >25% of the bone marrow.
6. Uncontrolled brain metastases. Patients with treated brain metastases (resection or radiotherapy) are eligible if brain metastases have responded to treatment as documented by CT or MRI scan obtained at >=2 weeks after completion of radiation therapy, neurologic symptoms are absent, and steroids have been discontinued.
7. Suspected, diffuse idiopathic interstitial lung disease or pulmonary fibrosis.
8. Diagnosis of second malignancy within the last 3 years (with the exception of carcinoma in situ of the cervix, squamous or basal cell skin cancer, thyroid cancer, ductal carcinoma in situ [DCIS], or lobular carcinoma in situ [LCIS]).
9. Any of the following <=12 months prior to starting study treatment:

   * myocardial infarction;
   * severe unstable angina;
   * congestive heart failure;
   * ongoing cardiac dysrhythmia.
10. Family history of idiopathic cardiomyopathy or uncontrolled heart arrhythmia.
11. Patients with previous allergy or hypersensitivity to anthracyclines.
12. Patients who have had a ≥10% drop in LVEF on previous anthracycline therapy.
13. Palliative radiotherapy to areas of metastatic breast cancer must have been completed >7 days prior to the first dose of study treatment. The exception is radiotherapy for brain metastases, which must be completed >=21 days prior to study treatment. (Note: Any measurable lesion that has been previously irradiated will not be considered as a target lesion).
14. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
15. History of seropositive HIV, or patients who are receiving immunosuppressive medications that increase the risk of neutropenic complications.
16. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
17. Use of any non-approved or investigational agent <=30 days of administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (16):
- United States (16):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Baptist Hospital East, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - Berks Hematology Oncology Associates, West Reading, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Peninsula Cancer Institute, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at multiple dose levels into the Dose Escalation (Phase I) portion of this study to determine the safest dose of this regime (MTD - Maximum Tolerated Dose). Upon determination of this dose, patients being treated at the MTD proceeded to the Dose Expansion (Phase II) portion of the study and additional patients were recruited
Groups:
- Dose Level 1: Amrubicin - 90 mg/m^2 by intravenous (IV) every 21 days
- Dose Level 2: Amrubicin - 100 mg/m^2 IV every 21 days
- Dose Level 3; Phase II: Amrubicin - 110 mg/m^2 IV every 21 days
- Dose Level 4: Amrubicin - 120 mg/m^2 every 21 days
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Phase II
Started | 3 | 3 | 3 | 6 | 63
Completed | 0 (Patients were on-study until determination of the Maximum Tolerated Dose (MTD)) | 0 (Patients were on-study until determination of the Maximum Tolerated Dose (MTD)) | 3 | 0 (Patients were on-study until determination of the Maximum Tolerated Dose (MTD)) | 0
Not Completed | 3 | 3 | 0 | 6 | 63

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Dose Level 1: Amrubicin -90 mg/m^2 by intravenous(IV) every 21days
- Phase I - Dose Level 2: Amrubicin -100 mg/m^2 IV every 21days
- Phase I - Dose Level 3; Phase II - Dose Level 3: Amrubicin -110 mg/m^2 IV every 21days
- Phase I - Dose Level 4: Amrubicin -120 mg/m^2 every 21 days
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3 | Phase I - Dose Level 4 | Phase II - Dose Level 3 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 63 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 6 | 44 | 58
  >=65 years | 0 | 1 | 0 | 0 | 19 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 6 | 63 | 78
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 3 | 4
  Not Hispanic or Latino | 1 | 1 | 3 | 5 | 53 | 63
  Unknown or Not Reported | 2 | 2 | 0 | 0 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 7 | 8
  White | 2 | 3 | 3 | 6 | 53 | 67
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) of MTD/Phase II Patients
Description: Progression-free survival is measured from Day 1 of study drug administration to disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death on the study. Progression is defined in RECIST v1.1 as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesions. This outcome measure is reported for all patients treated at the same dose level and is not separated into Phase I and Phase II. The phase I and phase II results are not separated as the timing of enrollment (early in phase 1 or later phase II) is not relevant to the outcome measure.
Time Frame: every 6 weeks until progressive disease
Population: Patients who received the dose level 3 MTD dose/Phase II dose (Amrubicin -110 mg/m^2) are included in the analysis. The 3, dose level 3 phase I pts and 63 phase II pts treated at this dose level are all combined to evaluate the efficacy of the MTD/phase II dose. The phase I and phase II results are not separated out as the timing of their enrollment (early in phase 1 or later phase II) is not relevant to the outcome measure. The other 12 phase I pts who were not treated at the MTD are excluded.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Amrubicin: Systemic therapy with amrubicin
Arm/Group | Amrubicin
Number analyzed (Participants) | 66
months | 4.0 [2.5 to 5.8]

2. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: Assessments will be made through analysis of the reported incidence of treatment-emergent Serious Adverse Events (SAEs) and non-serious adverse events (AEs).
Time Frame: every 6 weeks until treatment discontinuation, up to 43 months
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Amrubicin -90 mg/m^2 by intravenous(IV) every 21days
- Dose Level 2: Amrubicin -100 mg/m^2 IV every 21days
- Dose Level 3: Amrubicin -110 mg/m^2 IV every 21days
- Dose Level 4: Amrubicin -120 mg/m^2 IV every 21 days
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 66 | 6
Participants | 3 | 3 | 65 | 6

3. Secondary Outcome: Overall Survival (OS) of MTD/Phase II Patients
Description: Measured from Day 1 of study drug administration to date of death due to any cause. This outcome measure is reported for all patients treated at the same dose level and is not separated into Phase I and Phase II. The phase I and phase II results are not separated as the timing of enrollment (early in phase 1 or later phase II) is not relevant to this outcome measure.
Time Frame: every 6 weeks until treatment discontinuation, up to 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amrubicin
Number analyzed (Participants) | 66
months | 14.4 [10.1 to 18.5]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: The number of patients with observed complete response [CR] or partial response [PR]. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. This outcome measure is reported for all patients treated at the same dose level and is not separated into Phase I and Phase II. The phase I and phase II results are not separated as the timing of enrollment (early in phase 1 or later phase II) is not relevant to the outcome measure.
Time Frame: every 6 weeks until treatment discontinuation, up to 43 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Amrubicin
Number analyzed (Participants) | 66
participants | 12

ADVERSE EVENTS:
Time Frame: every 3 weeks up to 43 months
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from the day of the first dose to 30 days after the last dose of the study medication and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Groups:
- Dose Level 2: Amrubicin - 100 mg/m^2 by intravenous (IV) every 21 days
- Dose Level 3 (MTD)/Phase II: Amrubicin - 110 mg/m^2 by intravenous (IV) every 21 days Includes patients treated at the MTD in Dose Level 3 phase 1 and in phase II
- Dose Level 4: Amrubicin - 120 mg/m^2 by intravenous (IV) every 21 days
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 (MTD)/Phase II | Dose Level 4
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 5/66 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 65/66 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (MTD)/Phase II (N=66) | Dose Level 4 (N=6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PULMONARY INFILTERATES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (MTD)/Phase II (N=66) | Dose Level 4 (N=6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (9) | 0 (0)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 6 (17) | 0 (0)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 8 (39) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 32 (126) | 3 (6)
ANEMIA (Blood and lymphatic system disorders) | 1 (7) | 3 (12) | 27 (130) | 3 (5)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 2 (7) | 21 (40) | 3 (5)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (7) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 14 (39) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 6 (12) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (16) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 15 (49) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 6 (13) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 18 (48) | 1 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 9 (26) | 0 (0)
DECREASED BREATH SOUNDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (13) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (13) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 9 (24) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 12 (13) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 4 (9) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 10 (49) | 0 (0)
EDEMA (General disorders) | 0 (0) | 1 (4) | 7 (19) | 0 (0)
FATIGUE (General disorders) | 2 (5) | 2 (11) | 47 (203) | 4 (10)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 9 (16) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 8 (15) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (7) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (9) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (9) | 34 (83) | 3 (7)
MUCOSITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 9 (11) | 2 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (41) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (6) | 2 (9) | 25 (82) | 4 (5)
NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 11 (58) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (8) | 36 (87) | 5 (8)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (17) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 19 (49) | 5 (9)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (2)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 15 (26) | 2 (2)
WEIGHT LOSS (Investigations) | 0 (0) | 0 (0) | 6 (11) | 0 (0)
PAIN (General disorders) | 2 (3) | 2 (14) | 0 (0) | 4 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from the date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish results until 18 mos. after the trial has been completed at all sites.